CLINICAL TRIAL: NCT00111878
Title: Dose-Escalating Study to Evaluate MEDI-534 in Healthy Adults
Brief Title: Study to Evaluate MEDI-534 in Healthy Adults
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Other Study IDs: MI-CP119
Record Dates: First submitted 2005-05-26; First posted 2005-05-27 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2007-07

CONDITIONS: Respiratory Syncytial Virus Infections; Parainfluenza Infections
Keywords: Respiratory Syncytial Virus (RSV) and Parainfluenza Virus Type 3 (PIV3)
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: MEDI-534

SUMMARY:
The primary objective of this study is to describe the safety and tolerability of a single dose of MEDI-534 when administered to healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18 through 40 years (not yet reached their 41st birthday) on the day of randomization
* Healthy by medical history and physical examination
* Available by telephone
* Signed written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization obtained from the volunteer
* Sexually active females, unless surgically sterile or at least 1 year post-menopausal, must have used an effective method of avoiding pregnancy (including oral, implanted, or transdermal contraceptives, intrauterine device (IUD), female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for at least 30 days prior to dosing of study vaccine, and must agree to continue using such precautions for at least 30 days after dosing; the volunteer must also have a negative serum pregnancy test within 7 days prior to dosing of study vaccine and a negative urine pregnancy test on the day of study vaccine dosing prior to administration
* Sexually active males, unless surgically sterile, must use an effective method of birth control (condom or abstinence) and must agree to continue using such precautions for at least 30 days after dosing
* Ability to understand and comply with the requirements of the protocol as judged by the investigator
* Ability to complete the follow-up period of 6 months following dosing as required by the protocol

Exclusion Criteria:

* Acute illness on the day of randomization
* Fever (greater than or equal to 99.5°F oral or greater than or equal to 100.1°F tympanic) and/or respiratory illness (e.g., cough or sore throat) within 7 days prior to randomization
* Any drug therapy (chronic or other) within 7 days prior to randomization (except for certain medications such as contraceptives, topical [i.e., dermatologic] corticosteroids, or infrequent use of over-the-counter pain relievers, following approval from the sponsor) or expected receipt through 28 days after study vaccine dosing
* Receipt of immunoglobulin or blood products within 90 days prior to screening or expected receipt through 28 days after study vaccine dosing
* Receipt of any investigational drug within 60 days prior to randomization or expected receipt during the study period (i.e., through 180 days after study vaccine dosing)
* Receipt of an approved vaccine within 30 days prior to randomization or expected receipt through 28 days after study vaccine dosing
* History of immunodeficiency or receipt of immunosuppressive agents, or expected receipt of an immunosuppressive agent through 28 days after study vaccine dosing
* Close contact at home or in the workplace with children under 2 years of age
* Household contact who is immunocompromised; volunteer should also avoid close contact with immunocompromised individuals for at least 21 days after vaccination
* History of hypersensitivity to kanamycin or other aminoglycoside antibiotics (gentamicin, tobramycin, etc.)
* Previous medical history, or evidence, of an intercurrent or chronic illness that, in the opinion of the investigator, may compromise the safety of the volunteer
* Any evidence of end organ dysfunction
* Current, or history of, clinically significant abnormality on electrocardiogram (ECG) (screening ECG must be within 30 days prior to randomization)
* Evidence of active infection with HIV or hepatitis A, B, or C virus, or serologic evidence of past infection with hepatitis B or C virus
* At screening (must be within 7 days prior to randomization), any of the following laboratory tests outside of the laboratory normal range: CBC: hemoglobin (Hgb), WBC count, platelet count; AST, ALT, BUN, creatinine; or other abnormal laboratory value in the screening panel that, in the opinion of the principal investigator, may potentially confound analysis of study results
* Nursing mother
* History of alcohol or drug abuse in the past 2 years
* History of medical diagnosis of asthma, reactive airway disease, or chronic obstructive pulmonary disease (COPD)
* History of any smoking in the past 5 years
* Previous vaccination against Respiratory Syncytial Virus (RSV) or Parainfluenza Virus Type 3 (PIV3) in a clinical trial
* Employees of the research center, any individuals involved with the conduct of the study, or family members of such individuals
* Any condition that, in the opinion of the investigator, might interfere with study vaccine evaluation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120
Dates: Start 2005-04; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Gomez, MD, Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Children's Hospital, Columbus, Ohio
  - Primary Physicians Research, Pittsburgh, Pennsylvania
  - Radiant Research, Dallas, Texas